CLINICAL TRIAL: NCT06196398
Title: Effects of Medical Treatment of Intracranial Atherosclerotic Diseases Based on Magnetic Resonance Fractional Flow Reserve
Brief Title: Effects of Medical Treatment of ICAS With Hemodynamic Disorders Based on MR-FFR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: National Key Research and Development Project, China (Unknown)
Responsible Party: Sponsor
Other Study IDs: XWFFR-3
Record Dates: First submitted 2023-12-25; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Stroke, Ischemic; Intracranial Atherosclerosis
Keywords: Intracranial atherosclerotic diseases; Fractional Flow Reserve; Hemodynamics; Stroke
MeSH Terms: conditions — Ischemic Stroke; Intracranial Arteriosclerosis; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Decompensated blood flow reserve: ICAS patients with decompensated cerebral blood flow reserve diagnosed by MR-FFR (FFR baseline≥0.81).
  Interventions: Drug: Standard Medical Treatment on the basis of anti-platelet therapy
- Normal blood flow reserve: ICAS patients with normal cerebral blood flow reserve determined by MR-FFR (FFR baseline<0.81).
  Interventions: Drug: Standard Medical Treatment on the basis of anti-platelet therapy

INTERVENTIONS:
Drug: Standard Medical Treatment on the basis of anti-platelet therapy — 1. Anti-platelet therapy: aspirin 75mg+clopidogrel 100mg will be applied for patients with severe ICAS stenosis (70%-90%) suffering stroke or TIA within 30 days. After 90 days, single anti-platelet therapy will be continued.
  2. Intensive statin therapy: Statins with high doses
  3. Blood pressure: below 140/90mmHg
  4. LDL: less than 1.81mmol/L(70mg/dl)
  5. Fasting blood glucose controlled to 5.9mmol/L, and glycosylated hemoglobin A1c reduced to less than 7%
  6. Cigarette and alcohol quitting
  7. Oral anticoagulants for atrial fibrillation

SUMMARY:
This multicenter prospective cohort study aims to compare the difference in the effects of medical treatment within 1 year between the two groups of ICAS patients divided hemodynamically by Magnetic Resonance Fractional Flow Reserve. PC MRA will be applied for FFR measurement. The primary outcome is the composite of ischemic stroke or death related to the qualifying artery territory for 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged from 30 to 80 with symptomatic ICAS lesion in anterior circulation.
2. 50% to 99% stenosis (in accordance with modified WASID method) confirmed by DSA, CTA or MRA.
3. mRS 0-2 points
4. Informed of the study protocol and objectives.

Exclusion Criteria:

1. Previous endovascular treatment or surgery for cerebrovascular diseases
2. Large cerebral infarction (more than 1/2 MCA perfusion area) according to MRI
3. Combined with other neurological diseases, such as aneurysm, arteriovenous malformation, tumor, hydrocephalus, cerebral trauma, cerebral hemorrhage, multiple sclerosis, epilepsy and intracranial infection.
4. Pregnancy or in the preparation for pregnancy
5. Patients who cannot tolerate or do not allow MR screening, including metal implanting and claustrophobia
6. Contraindication for antiplatelet drugs or statins
7. Patients with severe dementia or mental disorders, who cannot cooperate with examination

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic, moderate to severe stenosis of major arteries in intracranial anterior circulation. The stenosis degree is ≥ 50%, confirmed by imaging evidence, according to modified WASID criteria.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
The composite of ischemic stroke or death related to the qualifying artery territory | 1 year

SECONDARY OUTCOMES:
Functional evaluation | 1 year
  Modified Rankin Scale score

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China